CLINICAL TRIAL: NCT05264207
Title: Nursing Students' Visits to Older Adults With Multiple Chronic Conditions: Effects on Self-care and Other Related Variables (VISITAME)
Brief Title: Nursing Students' Visits to Older Adults With Multiple Chronic Conditions
Acronym: VISITAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Jose Manuel Hernandez Padilla, Associate Professor (Profesor Titular), Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PID2020-117579RA-I00
Record Dates: First submitted 2022-02-14; First posted 2022-03-03 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Chronic Disease
Keywords: chronic disease; older adult; self-care; home-visit; nursing student
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Older adults who meet the inclusion criteria and voluntarily accept to participate in this study will be randomly allocated to one of two arms: intervention group (arm 1) or control group (arm 2). Participants from both arms will be assessed at the same time for data collection purposes (pre-test, post-test and 6-month follow-up) and they will be exposed to the experimental condition (intervention group) or the control condition (control group) at the same time for 12-weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The type of intervention on which the project is based does not allow for the participants to be masked and they will know to which group they are allocated. However, the team that will collect data (assessors) will not know the group to which each participant is allocated. To ensure assessor masking, participants will be instructed to never reveal the group to which they have been assigned and assessors will be instructed to never ask the participants to which group they have been assigned. The assessors will not participate in the recruitment process, the supervision of nursing students' home-visits, nor the data analysis process. The group to which the participants have been allocated will be numerically coded (not labelled) in the database and the researchers in charge of data analysis will not know which numerical code refers to the intervention group and which code refers to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants allocated to the 'intervention group' arm will receive the usual care offered by the Public Andalusian Healthcare Service in conjunction with a 12-week nursing students' home-visit programme.
  Interventions: Behavioral: Nursing students' home-visit programme; Behavioral: Standard care from Public Andalusian Health Service
- Control group (Active Comparator): Participants allocated to the 'control group' arm will only receive the usual care offered by the Public Andalusian Healthcare Service for 12 weeks.
  Interventions: Behavioral: Standard care from Public Andalusian Health Service

INTERVENTIONS:
Behavioral: Nursing students' home-visit programme — 12-week home-visit program conducted by nursing students. Participants will receive weekly 45-minute visits. The visits will aim to promote self-care behaviours and will focus on:
  1. Self-care of chronic conditions and medication management
  2. Healthy habits: physical activity and healthy eating
  3. Access to social support resources
  4. Patients' rights and autonomous decision-making
  The visits program will follow the WHO recommendations for the implementation of health promotion activities. All topics will be assigned 3 visits. In the first visit, the students will assess the participants' information needs and preferences in relation to the topic addressed and will provide generic information about it. In the second visit, the students will present individually-tailored information and will use individually-adapted strategies to convey such information. In the third visit, the student will explore the impact of the two previous visits and reinforce self-care behaviours.
  Arms: Intervention group
Behavioral: Standard care from Public Andalusian Health Service — Standard care offered by the Public Andalusian Health Service in its portfolio of services for older adults with multiple chronic conditions and complex health conditions. As part of these services, older adults with multiple chronic conditions receive generic, written information on healthy eating, adapted physical activity, abandonment of toxic habits, environmental safety and emotional management when they are first diagnosed with a chronic condition. The action plans or protocols established in the care processes aimed at older people with chronic multimnorbidity do not include periodic home visits.

SUMMARY:
BACKGROUND

The concurrence of multiple chronic conditions in older adults is associated with increased healthcare expenditure, increased hospital admissions, consultations and pharmaceutical expenditure. Having been diagnosed with multiple chronic conditions is associated with biopsychosocial health deterioration, worsening quality of life and increased mortality in older adults. Consequently, older adults with multiple chronic conditions present complex health statuses that require healthcare professional to focus on promoting health and independence through self-care.

Available evidence suggests that the implementation of programs with individualized interventions focused on health promotion could improve self-care and other related variables in older people with chronic conditions. In this regard, the World Health Organization recommends the implementation of community health promotion programs including at least 5 home-visits carried out by healthcare professionals to promote self-care, independence, and quality of life amongst older adults with chronic conditions. However, the evidence on the cost-effectiveness of such visiting programs is inconsistent, which makes it difficult to integrate them into the services offered by public-funded healthcare systems. In search of more effective interventions to improve self-care and other related variables amongst older adults with multiple chronic conditions, nursing student visits could be a valid, effective alternative. Some studies suggest that the implementation of periodic follow-up programs (visits or telephone calls) by nursing students not only improves their knowledge and attitudes in relation to the care of older adults, but they could also have a positive impact on patients.

STUDY'S HYPOTHESIS

A program of supervised visits carried out by nursing students will significantly improve self-care behaviors and other related variables amongst older adults with multiple chronic conditions.

AIM

The aim of the VISITAME project is to examine the short-term (12 weeks) and medium-term (6 months) effects of a nursing students' home-visit programme on self-care behaviors amongst older adults with multiple chronic conditions.

STUDY DESIGN

A parallel two-arm randomized controlled trial (RCT) will be carried out. Participants will be randomly assigned to either an intervention group (IG) or a control group (CG).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Having been diagnosed with more than one chronic condition.
* Living at home (community-dwelling).
* Signing the informed consent to participate in the study.

Exclusion Criteria:

* Having cognitive impairment (Pfeiffer test > 2 failures).
* Having been diagnosed with a psychiatric condition (for example: schizophrenia).
* Being a beneficiary of any of the services offered by the Fund of the Spanish National System for Autonomy and Support for Dependency.
* Being a beneficiary of private personal assistance to help with functional dependency.
* Participate in a program of similar nature from any public or private entities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 252 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in self-care behaviours | Changes from baseline to 3-month and 6-month follow-up
  Self-care in chronic illness inventory (SC-CII). The SC-CII will be used to measure the primary outcome of the study: 'self-care behaviours'. The SC-CII is a self-administered inventory, comprised of 20 items divided into 3 scales. The self-care maintenance scale is comprised of 8 items that measure, on a five-point Likert scale (1=never, 5=always), the frequency with which patients perform health-maintenance behaviors. The self-care monitoring scale is comprised of 5 items that measure, on a five-point Likert scale (1=never, 5=always), the frequency with which patients perform health-monitoring behaviors. The 'self-care management' scale is comprised of 7 items that measure, on a five-point Likert scale (1=not at all likely, 5=very likely), the probability for a patient to perform health-management behaviors. The scores of the three tools are calculated individually (between 0 and 100). Higher scores are indicative of better self-care.

SECONDARY OUTCOMES:
Change in self-efficacy in self-care | Changes from baseline to 3-month and 6-month follow-up
  The participants' self-efficacy in self-care will be assessed with the Self-Efficacy in Self-Care Scale (SESCS). The SESCS is comprised of 10 items that can be responded using a 5-point, Likert type scale (1=not confident; 5=extremely confident) and assess self-efficacy related to self-care maintenance, monitoring, and management in people diagnosed with chronic conditions. The participants' total scores will be standardised to range from 0-100, with higher scores indicating higher levels of self-efficacy.
Change in loneliness | Changes from baseline to 3-month and 6-month follow-up
  UCLA Loneliness Scale (UCLA). UCLA will be used to measure the variable 'loneliness'. This self-administered scale measures how often older people experience feelings of loneliness. The UCLA is comprised of 10 items to be answered using a 4-point Likert scale (1=I often feel this way, 4=I never feel this way). Lower scores are indicative of a greater feeling of loneliness. It is suggested that scores <20 points could indicate severe loneliness, while scores of 20-30 points could be indicative of moderate loneliness.
Change in perceived social support | Changes from baseline to 3-month and 6-month follow-up
  DUKE-UNK-11 questionnaire of perceived social support (DUKE-11). The DUKE-11 will be used to measure the variable 'perceived social support'. The DUKE-11 questionnaire is self-administered and measures perceived functional social support with 11 items divided into two dimensions: 'confidant support' and 'affective support'. All items have 5 response options in Likert format (1=as much as I want, 5=much less than I want) and allow participants to indicate the frequency with which they receive social support. Scores can range from 11-55 points. Scores >32 points indicate low perceived social support.
Change in funcional capacity for activities of daily living | Changes from baseline to 3-month and 6-month follow-up
  Barthel Index (BI). The BI will be used to measure the variable 'functional independence' to carry out the BADL. The BI is a unidimensional, hetero-administered questionnaire with 10 items measuring participants' independence for feeding, moving from chair to bed, doing personal toileting, getting on and off the toilet, bathing oneself, walking on a level surface or propelling a wheelchair, ascending and descending stairs, dressing and undressing, continence of bowels, and controlling bladder. The assessor can complete the questionnaire by direct observation or by interviewing the participant. The score can range from 0-100 (90 for people in wheelchairs) and the level of functional independence is determined by the score obtained: independent (100 points), mild dependency (≥ 60 points), moderate dependency (40-55 points), severe dependency (20-35 points), total dependency (< 20 points).
Change in nutritional status | Changes from baseline to 3-month and 6-month follow-up
  Nutritional status will be assessed using the Mini Nutritional Assessment (MNA). The MNA is comprised of 18 items divided in two sections: screening and assessment. The screening section is comprised of 6 items that assess and will yield a total screening score that can be interpreted: a score ≥ 12 indicates the person is well nourished, a score of 8-11 indicates the person is at risk of malnutrition, and a score ≤ 7 indicates the person is malnourished. When the person's score ≤ 11, it is recommended to complete the assessment section to determine the factors that could be affecting their nutritional status. The assessment section is comprised of 12 weighted items (0-2 points per item) that must be added to the screening score to calculate a total MNA score. A person with a total MNA score of 24-30 is considered to have a normal nutritional status, whereas people with a total MNA score of 17-23.5 is at risk of malnourishment and people with a total MNA score < 17 are malnourished.
Change in diet quality | Changes from baseline to 3-month and 6-month follow-up
  The participants' diet quality will be assessed using the Mediterranean Diet Adherence Screener (MEDAS). The MEDAS is comprised of 14 items that measure the degree of adherence to the typical Mediterranean dietary pattern. The MEDAS includes 12 questions on food consumption frequency and 2 questions on food intake habits considered typical of the Spanish Mediterranean diet. Each question is scored 0 or 1. A total score ≥ 9 indicates good adherence to the Mediterranean Diet.
Change in health-related quality of life | Changes from baseline to 3-month and 6-month follow-up
  SF-12 quality of life questionnaire (SF-12). The SF-12 questionnaire will be used to measure the variable 'quality of life'. The SF-12 is a self-administered questionnaire that measures health-related quality of life in 12 items. The SF-12 is the shortened version of the SF-36. The SF-12 response options follow a Likert-type scale that assesses intensity or frequency, depending on the item. The number of response options for each item ranges from three to six and the total score must be transformed from 0 to 100. Higher scores indicate better health-related quality of life.
Change in dignity | Changes from baseline to 3-month and 6-month follow-up
  Patient Dignity Inventory (PDI). The PDI will be used to measure the 'dignity' variable. The PDI is a self-administered instrument comprised of 25 items that are distributed in 3 dimensions: 'psychological and existential stress', 'physical symptoms and dependency' and 'social support'. Using a 5-point Likert scale (1=Not a problem, 5=Overwhelming problem), participants must respond to what degree certain situations related to dignity have been a problem or concern for them in the last few days. Higher scores indicate greater affectation in the participants' sense of dignity.
Change in personal autonomy | Changes from baseline to 3-month and 6-month follow-up
  Maastricht Personal Autonomy Questionnaire (MPAQ). The MPAQ is a self-administered questionnaire comprised of 16 items divided into 3 dimensions. The 'dilemmas' dimension (6 items) measures the frequency with which older people experience conflicts between what they want to do and what is best for their health (1=never; 5=very often). The 'degree of autonomy' dimension measures the impact of dilemmas on the participants' autonomy (1=Not at all; 5=Yes, completely). The dimension 'working on autonomy' (5 items) measures the efforts made by the participants to maintain personal autonomy (1=No, not at all; 5=Yes, I do everything possible),. The total score of each dimension is calculated by adding the score of all the items and dividing it by the total number of items. Higher scores indicate that people face dilemmas more often, experience a greater degree of autonomy, and work harder to maintain or achieve their autonomy.
Change in falls | Changes from baseline to 3-month and 6-month follow-up
  Number and place of falls in the last 6 months
Change in hospital admissions | Changes from baseline to 3-month and 6-month follow-up
  Number and cause of hospital admissions in the last 6 months
Change in visits to emergency departments | Changes from baseline to 3-month and 6-month follow-up
  Number and cause of visits to the emergency department in the last 6 months

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Hernández Padilla, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Universidad de Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared once the study is finalised and the main results are published. IPD can be obtained by contacting the responsible party (j.hernandez-padilla@ual.es)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Two years (24 months) after the study completion.
Access Criteria: The PI must be contacted and a minimum number of co-authors from the research team must be included in any publication

REFERENCES:
- [Background] Foguet-Boreu Q, Violan C, Rodriguez-Blanco T, Roso-Llorach A, Pons-Vigues M, Pujol-Ribera E, Cossio Gil Y, Valderas JM. Multimorbidity Patterns in Elderly Primary Health Care Patients in a South Mediterranean European Region: A Cluster Analysis. PLoS One. 2015 Nov 2;10(11):e0141155. doi: 10.1371/journal.pone.0141155. eCollection 2015. PMID 26524599
- [Background] Garin N, Olaya B, Perales J, Moneta MV, Miret M, Ayuso-Mateos JL, Haro JM. Multimorbidity patterns in a national representative sample of the Spanish adult population. PLoS One. 2014 Jan 20;9(1):e84794. doi: 10.1371/journal.pone.0084794. eCollection 2014. PMID 24465433
- [Background] Palladino R, Tayu Lee J, Ashworth M, Triassi M, Millett C. Associations between multimorbidity, healthcare utilisation and health status: evidence from 16 European countries. Age Ageing. 2016 May;45(3):431-5. doi: 10.1093/ageing/afw044. Epub 2016 Mar 24. PMID 27013499
- [Background] Picco L, Achilla E, Abdin E, Chong SA, Vaingankar JA, McCrone P, Chua HC, Heng D, Magadi H, Ng LL, Prince M, Subramaniam M. Economic burden of multimorbidity among older adults: impact on healthcare and societal costs. BMC Health Serv Res. 2016 May 10;16:173. doi: 10.1186/s12913-016-1421-7. PMID 27160080
- [Background] Laires PA, Perelman J. The current and projected burden of multimorbidity: a cross-sectional study in a Southern Europe population. Eur J Ageing. 2018 Sep 1;16(2):181-192. doi: 10.1007/s10433-018-0485-0. eCollection 2019 Jun. PMID 31139032
- [Background] Buja A, Rivera M, De Battisti E, Corti MC, Avossa F, Schievano E, Rigon S, Baldo V, Boccuzzo G, Ebell MH. Multimorbidity and Hospital Admissions in High-Need, High-Cost Elderly Patients. J Aging Health. 2020 Jun/Jul;32(5-6):259-268. doi: 10.1177/0898264318817091. Epub 2018 Dec 6. PMID 30522388
- [Background] McPhail SM. Multimorbidity in chronic disease: impact on health care resources and costs. Risk Manag Healthc Policy. 2016 Jul 5;9:143-56. doi: 10.2147/RMHP.S97248. eCollection 2016. PMID 27462182
- [Background] Bahler C, Huber CA, Brungger B, Reich O. Multimorbidity, health care utilization and costs in an elderly community-dwelling population: a claims data based observational study. BMC Health Serv Res. 2015 Jan 22;15:23. doi: 10.1186/s12913-015-0698-2. PMID 25609174
- [Background] Williams JS, Egede LE. The Association Between Multimorbidity and Quality of Life, Health Status and Functional Disability. Am J Med Sci. 2016 Jul;352(1):45-52. doi: 10.1016/j.amjms.2016.03.004. Epub 2016 Mar 18. PMID 27432034
- [Background] Gu J, Chao J, Chen W, Xu H, Zhang R, He T, Deng L. Multimorbidity and health-related quality of life among the community-dwelling elderly: A longitudinal study. Arch Gerontol Geriatr. 2018 Jan;74:133-140. doi: 10.1016/j.archger.2017.10.019. Epub 2017 Oct 28. PMID 29096228
- [Background] Bao XY, Xie YX, Zhang XX, Peng X, Huang JX, Du QF, Wang PX. The association between multimorbidity and health-related quality of life: a cross-sectional survey among community middle-aged and elderly residents in southern China. Health Qual Life Outcomes. 2019 Jun 24;17(1):107. doi: 10.1186/s12955-019-1175-0. PMID 31234889
- [Background] Makovski TT, Schmitz S, Zeegers MP, Stranges S, van den Akker M. Multimorbidity and quality of life: Systematic literature review and meta-analysis. Ageing Res Rev. 2019 Aug;53:100903. doi: 10.1016/j.arr.2019.04.005. Epub 2019 Apr 30. PMID 31048032
- [Background] Liu J, Yu W, Zhou J, Yang Y, Chen S, Wu S. Relationship between the Number of Noncommunicable Diseases and Health-Related Quality of Life in Chinese Older Adults: A Cross-Sectional Survey. Int J Environ Res Public Health. 2020 Jul 17;17(14):5150. doi: 10.3390/ijerph17145150. PMID 32708844
- [Background] Makovski TT, Le Coroller G, Putrik P, Choi YH, Zeegers MP, Stranges S, Ruiz Castell M, Huiart L, van den Akker M. Role of clinical, functional and social factors in the association between multimorbidity and quality of life: Findings from the Survey of Health, Ageing and Retirement in Europe (SHARE). PLoS One. 2020 Oct 20;15(10):e0240024. doi: 10.1371/journal.pone.0240024. eCollection 2020. PMID 33079931
- [Background] Nunes BP, Flores TR, Mielke GI, Thume E, Facchini LA. Multimorbidity and mortality in older adults: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2016 Nov-Dec;67:130-8. doi: 10.1016/j.archger.2016.07.008. Epub 2016 Aug 2. PMID 27500661
- [Background] Wei MY, Mukamal KJ. Multimorbidity and Mental Health-Related Quality of Life and Risk of Completed Suicide. J Am Geriatr Soc. 2019 Mar;67(3):511-519. doi: 10.1111/jgs.15678. Epub 2018 Nov 24. PMID 30471103
- [Background] Feng X, Tan X, Riley B, Zheng T, Bias T, Sambamoorthi U. Polypharmacy and Multimorbidity Among Medicaid Enrollees: A Multistate Analysis. Popul Health Manag. 2018 Apr;21(2):123-129. doi: 10.1089/pop.2017.0065. Epub 2017 Jul 6. PMID 28683221
- [Background] Nguyen TN, Ngangue P, Haggerty J, Bouhali T, Fortin M. Multimorbidity, polypharmacy and primary prevention in community-dwelling adults in Quebec: a cross-sectional study. Fam Pract. 2019 Nov 18;36(6):706-712. doi: 10.1093/fampra/cmz023. PMID 31104072
- [Background] Vetrano DL, Palmer K, Marengoni A, Marzetti E, Lattanzio F, Roller-Wirnsberger R, Lopez Samaniego L, Rodriguez-Manas L, Bernabei R, Onder G; Joint Action ADVANTAGE WP4 Group. Frailty and Multimorbidity: A Systematic Review and Meta-analysis. J Gerontol A Biol Sci Med Sci. 2019 Apr 23;74(5):659-666. doi: 10.1093/gerona/gly110. PMID 29726918
- [Background] Hanlon P, Nicholl BI, Jani BD, Lee D, McQueenie R, Mair FS. Frailty and pre-frailty in middle-aged and older adults and its association with multimorbidity and mortality: a prospective analysis of 493 737 UK Biobank participants. Lancet Public Health. 2018 Jul;3(7):e323-e332. doi: 10.1016/S2468-2667(18)30091-4. Epub 2018 Jun 14. PMID 29908859
- [Background] Kristensen K, Konig HH, Hajek A. The association of multimorbidity, loneliness, social exclusion and network size: findings from the population-based German Ageing Survey. BMC Public Health. 2019 Oct 28;19(1):1383. doi: 10.1186/s12889-019-7741-x. PMID 31660910
- [Background] Hajek A, Kretzler B, Konig HH. Multimorbidity, Loneliness, and Social Isolation. A Systematic Review. Int J Environ Res Public Health. 2020 Nov 23;17(22):8688. doi: 10.3390/ijerph17228688. PMID 33238506
- [Background] Kristensen K, Konig HH, Hajek A. The longitudinal association of multimorbidity on loneliness and network size: Findings from a population-based study. Int J Geriatr Psychiatry. 2019 Oct;34(10):1490-1497. doi: 10.1002/gps.5158. Epub 2019 Jun 25. PMID 31172559
- [Background] Stickley A, Koyanagi A. Physical multimorbidity and loneliness: A population-based study. PLoS One. 2018 Jan 24;13(1):e0191651. doi: 10.1371/journal.pone.0191651. eCollection 2018. PMID 29364978
- [Background] Kadambi S, Abdallah M, Loh KP. Multimorbidity, Function, and Cognition in Aging. Clin Geriatr Med. 2020 Nov;36(4):569-584. doi: 10.1016/j.cger.2020.06.002. Epub 2020 Aug 16. PMID 33010895
- [Background] Wang XX, Lin WQ, Chen XJ, Lin YY, Huang LL, Zhang SC, Wang PX. Multimorbidity associated with functional independence among community-dwelling older people: a cross-sectional study in Southern China. Health Qual Life Outcomes. 2017 Apr 17;15(1):73. doi: 10.1186/s12955-017-0635-7. PMID 28412945
- [Background] Bao J, Chua KC, Prina M, Prince M. Multimorbidity and care dependence in older adults: a longitudinal analysis of findings from the 10/66 study. BMC Public Health. 2019 May 16;19(1):585. doi: 10.1186/s12889-019-6961-4. PMID 31096943
- [Background] Wang C, Pu R, Li Z, Ji L, Li X, Ghose B, Huang R, Tang S. Subjective health and quality of life among elderly people living with chronic multimorbidity and difficulty in activities of daily living in rural South Africa. Clin Interv Aging. 2019 Jul 17;14:1285-1296. doi: 10.2147/CIA.S205734. eCollection 2019. PMID 31409978
- [Background] van Gennip IE, Pasman HR, Oosterveld-Vlug MG, Willems DL, Onwuteaka-Philipsen BD. The development of a model of dignity in illness based on qualitative interviews with seriously ill patients. Int J Nurs Stud. 2013 Aug;50(8):1080-9. doi: 10.1016/j.ijnurstu.2012.12.014. Epub 2013 Jan 8. PMID 23312465
- [Background] Ferretti, F., Pozza, A., Pallassini, M. et al. Gender invariance of dignity in non-terminal elderly patients with chronic diseases: a multicentric study. Qual Quant 53, 1645-1656 (2019). https://doi.org/10.1007/s11135-018-00831-z
- [Background] BLACK, K., & DOBBS, D. (2014). Community-dwelling older adults' perceptions of dignity: core meanings, challenges, supports and opportunities. Ageing and Society, 34(8), 1292-1313.
- [Background] Oosterveld-Vlug MG, Pasman HR, van Gennip IE, Muller MT, Willems DL, Onwuteaka-Philipsen BD. Dignity and the factors that influence it according to nursing home residents: a qualitative interview study. J Adv Nurs. 2014 Jan;70(1):97-106. doi: 10.1111/jan.12171. Epub 2013 May 26. PMID 23711199
- [Background] Wallace E, Salisbury C, Guthrie B, Lewis C, Fahey T, Smith SM. Managing patients with multimorbidity in primary care. BMJ. 2015 Jan 20;350:h176. doi: 10.1136/bmj.h176. No abstract available. PMID 25646760
- [Background] Riegel B, Jaarsma T, Stromberg A. A middle-range theory of self-care of chronic illness. ANS Adv Nurs Sci. 2012 Jul-Sep;35(3):194-204. doi: 10.1097/ANS.0b013e318261b1ba. PMID 22739426
- [Background] Doroszkiewicz H, Sierakowska M. Factors associated with risk of care dependency in disabled geriatric patients. Scand J Caring Sci. 2021 Mar;35(1):134-142. doi: 10.1111/scs.12827. Epub 2020 Feb 24. PMID 32091637
- [Background] Lommi M, Matarese M, Alvaro R, Piredda M, De Marinis MG. The experiences of self-care in community-dwelling older people: a meta-synthesis. Int J Nurs Stud. 2015 Dec;52(12):1854-67. doi: 10.1016/j.ijnurstu.2015.06.012. Epub 2015 Jul 17. PMID 26296653
- [Background] Lee E, Park E. Self-care behavior and related factors in older patients with uncontrolled hypertension. Contemp Nurse. 2017 Dec;53(6):607-621. doi: 10.1080/10376178.2017.1368401. Epub 2017 Aug 29. PMID 28831843
- [Background] Borhaninejad V, Shati M, Bhalla D, Iranpour A, Fadayevatan R. A Population-Based Survey to Determine Association of Perceived Social Support and Self-Efficacy With Self-Care Among Elderly With Diabetes Mellitus (Kerman City, Iran). Int J Aging Hum Dev. 2017 Dec;85(4):504-517. doi: 10.1177/0091415016689474. Epub 2017 Jan 24. PMID 28114826
- [Background] Mendoza-Nunez VM, Flores-Bello C, Correa-Munoz E, Retana-U Galde R, Ruiz-Ramos M. Relationship between social support networks and diabetes control and its impact on the quality of life in older community-dwelling Mexicans. Nutr Hosp. 2016 Nov 29;33(6):1312-1316. doi: 10.20960/nh.776. PMID 28000458
- [Background] Yang SO, Jeong GH, Kim SJ, Lee SH. Correlates of self-care behaviors among low-income elderly women with hypertension in South Korea. J Obstet Gynecol Neonatal Nurs. 2014 Jan-Feb;43(1):97-106. doi: 10.1111/1552-6909.12265. Epub 2013 Dec 19. PMID 24354464
- [Background] Buck HG, Dickson VV, Fida R, Riegel B, D'Agostino F, Alvaro R, Vellone E. Predictors of hospitalization and quality of life in heart failure: A model of comorbidity, self-efficacy and self-care. Int J Nurs Stud. 2015 Nov;52(11):1714-22. doi: 10.1016/j.ijnurstu.2015.06.018. Epub 2015 Jul 17. PMID 26234935
- [Background] Seid MA. Health-related quality of life and extent of self-care practice among heart failure patients in Ethiopia. Health Qual Life Outcomes. 2020 Feb 14;18(1):27. doi: 10.1186/s12955-020-01290-7. PMID 32059670
- [Background] Lee MK, Oh J. Health-Related Quality of Life in Older Adults: Its Association with Health Literacy, Self-Efficacy, Social Support, and Health-Promoting Behavior. Healthcare (Basel). 2020 Oct 16;8(4):407. doi: 10.3390/healthcare8040407. PMID 33081352
- [Background] Imaginario C, Rocha M, Machado P, Antunes C, Martins T. Self-care profiles of the elderly institutionalized in Elderly Care Centres. Arch Gerontol Geriatr. 2018 Sep-Oct;78:89-95. doi: 10.1016/j.archger.2018.05.012. Epub 2018 May 31. PMID 29935371
- [Background] Mlinac ME, Feng MC. Assessment of Activities of Daily Living, Self-Care, and Independence. Arch Clin Neuropsychol. 2016 Sep;31(6):506-16. doi: 10.1093/arclin/acw049. Epub 2016 Jul 29. PMID 27475282
- [Background] Chan EY, Samsudin SA, Lim YJ. Older patients' perception of engagement in functional self-care during hospitalization: A qualitative study. Geriatr Nurs. 2020 May-Jun;41(3):297-304. doi: 10.1016/j.gerinurse.2019.11.009. Epub 2019 Nov 29. PMID 31787364
- [Background] Xu X, Mishra GD, Jones M. Evidence on multimorbidity from definition to intervention: An overview of systematic reviews. Ageing Res Rev. 2017 Aug;37:53-68. doi: 10.1016/j.arr.2017.05.003. Epub 2017 May 13. PMID 28511964
- [Background] Weldring T, Smith SM. Patient-Reported Outcomes (PROs) and Patient-Reported Outcome Measures (PROMs). Health Serv Insights. 2013 Aug 4;6:61-8. doi: 10.4137/HSI.S11093. eCollection 2013. PMID 25114561
- [Background] Sasseville M, Chouinard MC, Fortin M. Patient-reported outcomes in multimorbidity intervention research: A scoping review. Int J Nurs Stud. 2018 Jan;77:145-153. doi: 10.1016/j.ijnurstu.2017.09.016. Epub 2017 Sep 29. PMID 29080440
- [Background] Black N. Patient reported outcome measures could help transform healthcare. BMJ. 2013 Jan 28;346:f167. doi: 10.1136/bmj.f167. PMID 23358487
- [Background] Lee HJ, Lee M, Ha JH, Lee Y, Yun J. Effects of healthcare interventions on psychosocial factors of patients with multimorbidity: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2020 Nov/Dec;91:104241. doi: 10.1016/j.archger.2020.104241. Epub 2020 Aug 25. PMID 32882587
- [Background] Poitras ME, Maltais ME, Bestard-Denomme L, Stewart M, Fortin M. What are the effective elements in patient-centered and multimorbidity care? A scoping review. BMC Health Serv Res. 2018 Jun 14;18(1):446. doi: 10.1186/s12913-018-3213-8. PMID 29898713
- [Background] World Health Organization. 2015. World report on aging and health. Available in URL: https://apps.who.int/iris/bitstream/handle/10665/186463/9789240694811_eng.pdf?sequence=1
- [Background] Brettschneider C, Luck T, Fleischer S, Roling G, Beutner K, Luppa M, Behrens J, Riedel-Heller SG, Konig HH. Cost-utility analysis of a preventive home visit program for older adults in Germany. BMC Health Serv Res. 2015 Apr 3;15:141. doi: 10.1186/s12913-015-0817-0. PMID 25884452
- [Background] Ruiz S, Snyder LP, Rotondo C, Cross-Barnet C, Colligan EM, Giuriceo K. Innovative Home Visit Models Associated With Reductions In Costs, Hospitalizations, And Emergency Department Use. Health Aff (Millwood). 2017 Mar 1;36(3):425-432. doi: 10.1377/hlthaff.2016.1305. PMID 28264943
- [Background] Tappenden P, Campbell F, Rawdin A, Wong R, Kalita N. The clinical effectiveness and cost-effectiveness of home-based, nurse-led health promotion for older people: a systematic review. Health Technol Assess. 2012;16(20):1-72. doi: 10.3310/hta16200. PMID 22490205
- [Background] Goehner A, Kricheldorff C, Bitzer EM. Trained volunteers to support chronically ill, multimorbid elderly between hospital and domesticity - a systematic review of one-on-one-intervention types, effects, and underlying training concepts. BMC Geriatr. 2019 May 2;19(1):126. doi: 10.1186/s12877-019-1130-2. PMID 31046693
- [Background] Knecht JG, Fischer B. Undergraduate Nursing Students' Experience of Service-Learning: A Phenomenological Study. J Nurs Educ. 2015 Jul;54(7):378-84. doi: 10.3928/01484834-20150617-04. PMID 26155029
- [Background] Davis RL, Beel-Bates C, Jensen S. The Longitudinal Elder Initiative: helping students learn to care for older adults. J Nurs Educ. 2008 Apr;47(4):179-82. doi: 10.3928/01484834-20080401-09. PMID 18468295
- [Background] Kruger BJ, Roush C, Olinzock BJ, Bloom K. Engaging nursing students in a long-term relationship with a home-base community. J Nurs Educ. 2010 Jan;49(1):10-6. doi: 10.3928/01484834-20090828-07. Epub 2010 Jan 4. PMID 19731887
- [Background] Conti G, Bowers C, O'Connell MB, Bruer S, Bugdalski-Stutrud C, Smith G, Bickes J, Mendez J. Examining the effects of an experiential interprofessional education activity with older adults. J Interprof Care. 2016;30(2):184-90. doi: 10.3109/13561820.2015.1092428. Epub 2016 Feb 25. PMID 26913632
- [Background] Walton J, Blossom H. The experience of nursing students visiting older adults living in rural communities. J Prof Nurs. 2013 Jul-Aug;29(4):240-51. doi: 10.1016/j.profnurs.2012.05.010. PMID 23910926
- [Background] Wheeler EC, Waterhouse JK. Telephone interventions by nursing students: improving outcomes for heart failure patients in the community. J Community Health Nurs. 2006 Fall;23(3):137-46. doi: 10.1207/s15327655jchn2303_1. PMID 16863399
- [Background] Ng KYY, Leung GYC, Tey AJ, Chaung JQ, Lee SM, Soundararajan A, Yow KS, Ngiam NHW, Lau TC, Wong SF, Wong CH, Koh GC. Bridging the intergenerational gap: the outcomes of a student-initiated, longitudinal, inter-professional, inter-generational home visit program. BMC Med Educ. 2020 May 11;20(1):148. doi: 10.1186/s12909-020-02064-x. PMID 32393249